CLINICAL TRIAL: NCT03733600
Title: Evaluation of the Xen Implant in Glaucoma Surgery
Acronym: Xen
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: XEN
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma: All patients followed for either early or moderate forms of primary or secondary open-angle glaucoma who had undergone surgery for Xen alone or in combination with cataract surgery for phacoemulisation of the lens.

SUMMARY:
Glaucoma is a blinding optic neuropathy that affects 60 million people around the world. Primary open-angle glaucoma is the most common etiology. The therapeutic arsenal now includes medicated hypotonic treatments, lasers and surgery. The most common glaucoma surgery in France is trabeculectomy and non-perforating deep sclerectomy. These are two filtering surgeries whose principle is to lower the intraocular pressure by creating a way of evacuation of the aqueous humor from the anterior chamber of the eye to the space sub conjunctival creating a bubble of filtration. The short-term complications with these techniques are early hypotonia and its attendant complications (choroidal detachment, maculopathy of hypotonia, haemorrhage...). In the medium term, blood pressure with deep anterior chamber, testify to a scleral flap too tight which may require suture lysis. Finally, the problems of excessive conjunctivo-tenon healing affect 25 to 30% of operated and are responsible for the majority of late blood pressure. In the longer term, the most common complication is cataracts. It can be complicated by a very serious endophthalmitis. A new minimally invasive therapeutic option has been developed that limits per and postoperative complications. In contrast to traditional techniques that have an ab externo approach, the ab interno approach of the proposed new technique involves the implantation of a collagen tube 6 mm in length and 45 μm of light called Xen® through the anterior chamber. This surgery can be performed alone or at the same time as a cataract surgery. The geometry of the Xen® implant has been studied to prevent major hypotonia. This new technique would also avoid the complications associated with conjunctival dissection, while being faster. A Xen® implant is nowadays indicated for simple surgery or combined with cataract surgery for open-angle, early-to-moderate, cataract and non-cataract glaucoma, progressive and unbalanced under local hypotonism therapy. Since June 2017, the Xen® technique is part of the routine at GhPSJ.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of surgery with Xen® implantation on intra-ocular pression drop in patients with primary or secondary open-angle glaucoma, beginner to moderate. The study will be proposed to all eligible patients operated between June 2017 and June 2018. After patient's non opposition, clinical data will be collected from patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for either early or moderate forms of primary or secondary open-angle glaucoma who had undergone surgery for Xen® alone or in combination with cataract surgery for phacoemulisation of the lens
* Patients operated between June 2017 and June 2018

Exclusion Criteria:

* Patient objecting to participate in the study
* Patient with other associated ophthalmological disease, except simple cataract already operated or operated simultaneously with the Xen® break without per or postoperative complication
* History of filter surgery, history of vitrectomy
* Close angle glaucoma
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient, operated between June 2017 and June 2018, followed for either early or moderate forms of primary or secondary open-angle glaucoma who had undergone surgery for Xen® alone or in combination with cataract surgery for phacoemulisation of the lens.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficiency of surgery with Xen | year 1
  The success of surgery will be evaluate with the intra-ocular pressure's measurement. Complete success corresponds to Intra-ocular pressure between 5 and 18 mmHg, with a relative decrease of more than 20% compared to the initial intra-ocular pressure, without having resorted to hypotonic treatments. Partial success corresponds to intra-ocular pressure between 5 and 18 mmHg but with an intra-ocular pressure reduction of less than 20% or with maintenance of a hypotonizing treatment. Therapeutic failure is defined as an intra-ocular pressure strictly greater than 18 mmHg or less than 5 mmHg.

SECONDARY OUTCOMES:
Evaluation of visual activity | year 1
  Visual acuity will be measure and compare to the preoperative visit to evaluate the efficiency of Xen.
Evaluation of visual fieldwill | year 1
  The visual fieldwill be measure and compare to the preoperative visit in order to evaluate the Xen's efficiency.
Measurement of Optic nerve excavation | year 1
  Optic nerve excavation will be measure and compare to the preoperative visit in order to evaluate of the efficiency of Xen.
Evaluation of the efficiency of Xen | year 1
  Number of hypotonizing drugs will be collecte and compare to the preoperative visit to evaluate yhe efficiency of Xen.
Evaluation of post-operative complications | year 1
  Post-operative complications will be collected.
Evaluation of reintervention rate | year 1
  Reintervention number will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Yves P LACHKAR, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided